CLINICAL TRIAL: NCT05269589
Title: Impact of a Home-based Heat Therapy Intervention on Markers of Cardiometabolic Function in Adults with Type 2 Diabetes
Brief Title: Home-based Heat Therapy for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Daniel Gagnon, Principal Investigator, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-2959
Record Dates: First submitted 2022-02-07; First posted 2022-03-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; Heat Exposure
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thermoneutral (Sham Comparator): Participants will immerse their feet in a foot bath with water maintained at 36°C
  Interventions: Other: Thermoneutral water
- Heat (Experimental): Participants will immerse their feet in a foot bath with water maintained at 42°C
  Interventions: Other: Hot water

INTERVENTIONS:
Other: Thermoneutral water — Participants will immerse their feet in a foot bath that contains thermoneutral water
  Arms: Thermoneutral
Other: Hot water — Participants will immerse their feet in a foot bath that contains hot water
  Arms: Heat

SUMMARY:
Insulin resistance and hyperglycemia predispose individuals with type 2 diabetes mellitus (T2DM) to endothelial dysfunction and a greater risk of cardiovascular diseases (CVD). Increased CVD risk in individuals with T2DM persists despite optimal pharmacological therapy, highlighting the need to identify complementary lifestyle interventions that improve cardiometabolic functions in this population. Evidence from animal models suggests that heat exposure improves metabolic functions. Notably, weekly heat exposure for 16 weeks blunts hyperinsulinemia and hyperglycemia induced by a high fat diet in mice. In parallel, studies in humans have shown that heat exposure improves vascular endothelial function. Based on such findings, it has been suggested that heat therapy may represent an effective lifestyle intervention to improve cardiometabolic functions. However, only 1 study has examined the impact of a heat therapy intervention on individuals with T2DM, demonstrating that 6 weeks of heat exposure reduces fasting plasma glucose and hemoglobin A1C. No study has considered potential vascular benefits of heat therapy in individuals with T2DM.

This project will investigate cardiometabolic responses to repeated heat exposure in men and women with T2DM. We will test the hypothesis that 12 weeks of heat therapy improves postprandial fatty acid handling, insulin sensitivity and endothelial function in individuals with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years
* Diagnosis of type 2 diabetes mellitus ≥1 year
* Stable medication ≥12 weeks

Exclusion Criteria:

* Class 3 obesity
* Hypertension not controled by medication
* Diagnosis of cardiac, renal and/or pulmonary disease
* Diagnosis of severe neuropathy and/or retinopathy
* Insulin therapy
* Fasting plasma triglycerides >5.0 mmol/L
* Fasting total cholesterol >7 mmol/l

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | Change from baseline to 12 weeks

SECONDARY OUTCOMES:
Insulin resistance (HOMA-IR) | Change from baseline to 12 weeks
Postprandial metabolism following meal | Change from baseline to 12 weeks
  Quantified over a 6-hour period following the ingestion of a standardized liquid meal
Peripheral endothelial function | Change from baseline to 12 weeks
  Brachial artery flow-mediated dilation
Post-occlusion reactive hyperemia | Change from baseline to 12 weeks
  Reactive hyperemia following 5 minutes of forearm ischemia
Ischemic handgrip exercise | Change from baseline to 12 weeks
  Reactive hyperemia following ischemic handgrip exercise
Arterial stiffness | Change from baseline to 12 weeks
  Carotid-femoral pulse wave velocity
Blood pressure | Change from baseline to 12 weeks
  24-hour ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Centre ÉPIC, Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No